CLINICAL TRIAL: NCT04288609
Title: Effectiveness of a Cognitive Remediation Intervention Based on Virtual Reality for Promotion of Cognitive Functioning and Participation in Daily Life Among Persons With Affective Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Geha Mental Health Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Geha Mental Health Center
Record Dates: First submitted 2020-02-10; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Affective Disorder
Keywords: affective disorder
MeSH Terms: conditions — Mood Disorders | interventions — Paper

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intendu FBT inpatient (Experimental): Motion Based Cognitive Video Games Software
  Interventions: Other: Intendu
- paper and pencil tasks (Active Comparator): paper and pencil tasks
  Interventions: Other: Paper and Pencil cognitive remediation training

INTERVENTIONS:
Other: Intendu — Cognitive remediation using VR adaptive platform for response inhibition, self-initiation, cognitive flexibility, sustained attention, divided attention, working memory, planning, persistence.
  Other Names: Motion Based Cognitive Video Games Software
  Arms: Intendu FBT inpatient
Other: Paper and Pencil cognitive remediation training — Cognitive remediation using paper and pencil tasks for response inhibition, self-initiation, cognitive flexibility, sustained attention, divided attention, working memory, planning, persistence.
  Other Names: Low-Tech remedial training
  Arms: paper and pencil tasks

SUMMARY:
The purpose of this study is to test the efficacy of remedial cognitive intervention using The Functional Brain Trainer VR (FBT, Intendo ©) to improve cognitive functioning, participation in daily life occupations, and functional capacity in the field of IADL among people with affective disorders receiving inpatient and daycare mental-health services.

DETAILED DESCRIPTION:
This study is an experimental study, in a pre-post design with a control group, the sampling is convenience. The study will include 40 people aged 18-60 with a diagnosis of Affective disorder based on DSM-5.

Inclusion criteria: age 18-60, Diagnosis of Major Depression or Bipolar disorder based on DSM-5; Mood stabilizing medication for at least 2 weeks, Exclusion criteria: Neurological disorders and neurodevelopmental conditions in addition to mental health diagnosis; Physical disability in addition to mental health conditions; Psychotic state; active substance abuse; custodian.

They will be recruited from active inpatient and daycare wards of the "Geha Mental Health Center", Israel and will be randomly allocated into two groups: experimental and control. An experimental group will attend 6 VR based cognitive remediation sessions of 30 minutes for training response inhibition, self-initiation, cognitive flexibility, sustained attention, divided attention, working memory, planning, persistence. The control group will complete 6 sessions of 30 minutes of low-tech (paper and pencil tasks) remedial training of the same cognitive components. These in addition to routine care. The evaluation for symptoms severity, cognition, functional capacity and participation in daily life activities will be conducted at the beginning of the study and after about 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60,
* Diagnosis of Major Depression or Bipolar disorder based on DSM-5;
* Mood stabilizing medication for at least 2 weeks,

Exclusion Criteria:

* Neurological disorders and neuro-developmental conditions in addition to mental health diagnosis;
* Physical disability in addition to mental health conditions;
* Psychotic state;
* active substance abuse;
* custodian

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
The Observed Tasks of Daily Living - Revised | 3 weeks
  Assessment of Functional capacity, score range 1 (dependent in the performance of daily life activities) up to 26 (fully independent in the performance of the daily life activities)
Adults Subjective Assessment of Participation | 3 weeks
  Questionnaire for assessment of participation in daily life activities: number of participated activities (from 1 to 52, the higher number indicates higher number of participated activities) and frequency of the participation (range from 1 indicates low frequency of participation up to 7 - higher frequency of the participation)

SECONDARY OUTCOMES:
The Neurobehavioral Cognitive Status Examination | 3 weeks
  Examination cognitive components of attention language, spatial skills, memory, calculations and reasoning. The score range for different sub-tests from 1 up to 4, 6, 8 or 12, with higher score indicates better cognitive functioning
Trail Making Test A & B | 3 weeks
  Measure of cognitive flexibility and psycho-motor processing speed, the score is a time needed for the test completion, less time that needed indicates better cognitive functioning
Category Fluency Test | 3 weeks
  Assessment of language fluency, the score is a number of produced words, the higher the number, the better cognitive fluency
Hamilton Depression Rating Scale Questionnaire | 3 weeks
  Assessment of the depressive symptoms, the higher score indicates more severe depressive symptoms.